CLINICAL TRIAL: NCT01279005
Title: Risk Taking Behaviour in MSM and the Denial of Sexually Transmitted Diseases and HIV - Focus Groups, Observational Study
Brief Title: Risk Taking Behaviour in MSM and the Denial of Sexually Transmitted Diseases and HIV
Acronym: MSM HIV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: NGO Via Libre (Other)
Responsible Party: Dr. Margalit Lorber, Rambam Medical Center, Haifa
Other Study IDs: 0425-10CTIL
Record Dates: First submitted 2011-01-09; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: MSM; HIV Infections; Risky Behaviors
Keywords: MSM; focus group; HIV; risk-taking; risk-denial; signature on inform consent, willing to participate, MSM either HIV positive or negative, age 20-50 years old
MeSH Terms: conditions — HIV Infections; Risk-Taking

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20-50 YEARS OLD MSM

SUMMARY:
Four focus groups , each of 10-15 males, ages 20-50 years old, MSM will be conducted by a medical sociologist. Two groups will be HIV negative participants and two groups of HIV positive MSM. Every group will meet for two hours. The focus group will be recorded and the collected data will be processed further for evaluation and extraction of the relevant information.

The volunteers will sign an inform consent prior to entrance to the study.

DETAILED DESCRIPTION:
The questions that will be discussed during the focus groups: The first sexual contact with a male, what is risk, risk taking behavior, control over your daily life, self esteem and evaluation, risk denial.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50
* MSM, willing to participate
* Agree to sign an inform consent

Exclusion Criteria:

* No exclusion criteria

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40-50 years old MSM
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-07 (Estimated)